CLINICAL TRIAL: NCT06699134
Title: Evaluation of Hi-Fatigue G Bone Cement With Gentamicin A Retrospective Data Collection
Brief Title: Hi-Fatigue G Bone Cement Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CME2020-38C
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Total Hip and Knee Arthroplasties
Keywords: Bone Cement; Knee Arthroplasty; Hip Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Patients with TKA: Patients with primary total knee replacement using Hi-Fatigue G Bone Cement and a Zimmer Biomet implant
  Interventions: Device: Total knee arthroplasty
- Patients with THA: Patients with primary total hip replacement using Hi-Fatigue G Bone Cement and a Zimmer Biomet implant
  Interventions: Device: Total Hip arthroplasty

INTERVENTIONS:
Device: Total knee arthroplasty — Primary total knee replacement using Hi-Fatigue G Bone Cement and a Zimmer Biomet implant
  Groups: Patients with TKA
Device: Total Hip arthroplasty — Primary total hip replacement using Hi-Fatigue G Bone Cement and a Zimmer Biomet implant
  Groups: Patients with THA

SUMMARY:
The objective of this retrospective monocentric study is to collect survivorship and clinical data confirming safety, performance and clinical benefits for the Hi-Fatigue G Bone Cement.

The assessments will include:

* Radiological analysis performed at different time points according to the standard of care of the hospital
* Implant survivorship and safety based on removal of a study device
* Patient reported outcome measures (PROMs)

Primary endpoint:

Assessment of radiolucent lines around the components (tibial, femoral, acetabular) at 5 years (in accordance with the hospital standard of care).

Secondary endpoints:

* Evaluation of implant survivorship and safety by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.
* Evaluation of PROMs
* Obtain information regarding the cementing technique and handling of the cement, if available

ELIGIBILITY:
Inclusion Criteria:

* Subject qualified for cemented TKA or THA with a Zimmer Biomet implant
* Subject is willing and able to give written informed consent for retrospective data collection and undergo interim and final evaluation (X-Ray & Scores completion)
* Subject > 18 years old

Exclusion Criteria:

* Muscle wasting
* Neuromuscular compromise in the affected limb
* Known hypersensitivity to any of the cement constituents
* Subjects with severe renal failure
* Bilateral interventions
* Subject is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, known alcohol or drug abuser, anticipated to be non-compliant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated with primary total knee or hip replacement using Hi-Fatigue G Bone Cement, a Zimmer Biomet implant, and who meet the inclusion / exclusion criteria for study participation.
  Two consecutive groups of patients that underwent cemented TKA or THA according to the instructions for use of both the respective implant and of Hi-Fatigue G Bone Cement.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Radiographic evaluation | From enrollment to the 5 year post-op follow up.
  Detection of radiolucent lines around the implant components (tibial, femoral, acetabular) at 5 years (in accordance with the hospital standard of care).

SECONDARY OUTCOMES:
Survivorship | From enrollment to the 5 year post-op follow up.
  Evaluation of implant survivorship and safety by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.
Patient reported outcome measures (PROM) | From enrollment to the 5 year post-op follow up.
  Evaluation of PROMs, collected in accordance with the hospital standard of care.
Cement Information | From enrollment to the 5 year post-op follow up.
  Obtain information regarding the cementing technique and handling of the cement, if available

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikum Weiden, Weiden, Bavaria, Germany